CLINICAL TRIAL: NCT06017024
Title: Evaluation of a New Microprocessor-Controlled Prosthetic Knee : A Prospective, Multicentered, Randomized Cross-over Trial
Brief Title: New Microprocessor-Controlled Prosthetic Knee Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Proteor Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A01266-37
Record Dates: First submitted 2023-07-19; First posted 2023-08-30 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: Micro-processor controlled knee; Lower Limb prosthesis; Patient-specific Functional Scale
MeSH Terms: conditions — Wounds and Injuries | interventions — Physical Examination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Current microprocessor-controlled knee (MPK) then New MPK (Experimental): Start using current MPK for 4 weeks before fitting new MPK and use it for 4 weeks
  Interventions: Device: microprocessor-controlled knee (MPK) assessment
- New MPK then Current MPK (Experimental): Start using new MPK for 4 weeks before fitting back current MPK and use it for 4 weeks
  Interventions: Device: microprocessor-controlled knee (MPK) assessment

INTERVENTIONS:
Device: microprocessor-controlled knee (MPK) assessment — The subject will wear the microprocessor-controlled knee prosthesis for 4 weeks, and then reply questionnaires and achieve functional tests

SUMMARY:
The target of this clinical investigation is to compare the achievement of personal functional goals using a new MPK and current MPK. Subjects will also run functional tests and questionnaires to compare performances and feedback with each prosthetic knee.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent
* Man or woman, more than 18 y.o
* Lower limb amputee KD or AKA, unilateral or bilateral
* K3/K4 activity level
* Already fitted with FR-reimbursed MPK
* Being comfortable in their socket (SCS>=5)

Exclusion Criteria:

* Protected person
* Pregnant or breast feeding lady
* Person having pathologies affecting their sensitivity
* Using walking aids
* Weighting more than 136kg
* Insufficient hip joint or pelvic voluntary muscle control
* Insufficient cognitive ability to charge the knee and care for the device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Personal goal achievement | test sessions 1 and 2 (20 minutes)
  Patient-specific Functional Scale - PSFS - [0-10], the higher the better

SECONDARY OUTCOMES:
Functional walking test - mobility capacity | test sessions 1 and 2 (8 minutes)
  6-minute walk test (6MWT)
Functional walking test - fast walking speed | test sessions 1 and 2 (1 minute)
  10-meter walk test (10mWT)
Functional test - ability to walk downhill | test sessions 1 and 2 (3 minutes)
  Hill assessment index (HAI) [0-11], the higher the better
Functional test - ability to walk downstairs | test sessions 1 and 2 (3 minutes)
  Stairs assessment index (SAI) [0-13], the higher the better
Questionnaire to assess comfort in the socket | test sessions 1 and 2 (1 minute)
  Socket comfort score (SCS) [0-10], the higher the better
Questionnaire to assess satisfaction | test sessions 1 and 2 (5 minutes)
  Quebec User Evaluation of Satisfaction with assistive Technology (QUEST = ESAT in French); the higher the better
Questionnaires to assess quality of life | test sessions 1 and 2 (5 minutes)
  Short Form (36) health survey (SF-36); the higher the better
Prosthesis Evaluation Questionnaire | test sessions 1 and 2 (29 minutes)
  PEQ, 8 sub-scales [0-100], the higher the better

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Léon Bérard, Hyères
  - Clinique du Dr Ster, Lamalou-les-Bains
  - UGECAM Nord-Est IRR, Nancy
  - Centre Mutualiste de Kerpape, Ploemeur
  - UGECAM La Tourmaline, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT06017024/SAP_000.pdf